CLINICAL TRIAL: NCT00261079
Title: The Evaluation of Efficacy and Safety of Fexofenadine 180mg Tablets for 7 Days in the Treatment of Pruritic Skin Disease
Brief Title: Fexofenadine in Pruritic Skin Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M016455_4125
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus | interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fexofenadine

SUMMARY:
Primary objective:

* To compare the efficacy and safety profile of Fexofenadine 180mg tablets plus prednicarbate(2.5mg/g) vs prednicarbate(2.5mg/g) alone in the treatment of pruritic skin disease

Secondary objective:

* To evaluate patient's satisfaction of Allegra treatment

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Main criteria are listed hereafter:

Inclusion Criteria:

* All patients diagnosed with atopic dermatitis, contact dermatitis

Exclusion Criteria:

* Other skin disease except atopic dermatitis, contact dermatitis.
* Subjects taken steroid within 4 weeks and antihistamine within 1 week before screening day.
* Pruritus localized only head and face
* Subjects with severe hepatic, renal, heart dysfunction.
* Subjects with history of alcohol and drug abuse.
* Pregnant and lactating women.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2005-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The change of physician's assessment on pruritic score before and after 7-day treatment.

SECONDARY OUTCOMES:
Patient visual analogue scale change and Overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Hyou-Young Rhim, MD, Study Director — Handok Inc.
Locations (1):
- Handok, Seoul, South Korea